CLINICAL TRIAL: NCT03666195
Title: Anti-Microbial Effect of Titanium Dioxide Nano Particles Incorporated Acrylic Resin Denture Base Materials in Completely Edentulous Patients: A Randomized Controlled Trial
Brief Title: The Anti-microbial Effect of Titanium Dioxide Nano Particles in Complete Dentures Made for Edentulous Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Ibrahim Badran, Teaching Asisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Mona's Protocol
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Candida Infection; Denture Stomatitis
Keywords: Nanoparticles; Titanium dioxide; biofilm; self cleansing; denture plaque; anti microbial
MeSH Terms: conditions — Candidiasis; Stomatitis, Denture

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessor will be blinded as well as the statistician and the participant.
  The outcome assessor will count the bacterial colony forming units without knowing the type of the denture material used (Conventional acrylic resin or acrylic resin modified by titanium dioxide nanoparticles)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): complete dentures will be fabricated using poly methyl methacrylate resin denture base material modified with 5%wt titanium dioxide nanoparticles.
  Interventions: Combination Product: Titanium Dioxide Nanoparticles
- Group B (No Intervention): complete dentures will be fabricated with poly methyl methacrylate resin denture base material.

INTERVENTIONS:
Combination Product: Titanium Dioxide Nanoparticles — incorporating titanium dioxide nanoparticles to PMMA, significantly decreases porosities in the denture resin, rendering titanium dioxide nanoparticles a suitable additive to denture base materials, as it also exhibits anti-microbial effects
  Other Names: Ultra fine titanium dioxide; TiO2
  Arms: Group A

SUMMARY:
Although cleaning dentures by immersion in chemical denture cleaning solutions is effective in reducing the number of bacteria, a large number remains adhering to the denture surface. Thus, the mechanical cleansing of dentures is imperative to remove adherent microbes, and prevent diseases. This is not always easy to achieve, due to un-compliant patients, or patients with diminished manual dexterity (e.g. Mani phalanx dysfunction or Rheumatoid Arthritis) that often require assistance in cleaning their dentures, which may not always be available.

Therefore, the modification of denture base materials to provide them with antibacterial properties to control oral biofilm formation, and producing dentures that can be cleaned by simply rinsing in water would prove to be valuable in oral hygienic management in complete denture-wearing patients.

DETAILED DESCRIPTION:
Nanoparticulate Metals as Antimicrobial Agents Many of the major medical breakthroughs in history, have been largely dependent on the antimicrobial effects of different metals. Mercury has been used medicinally in the treatment of syphilis, and skin diseases as far back as the 10th century in Europe, and 2nd Century BC in China. And till this day organomercurial compounds remain in use for their antiseptic, and disinfectant properties. Metals such as copper and zinc are now incorporated in micron size, in products such as toothpastes, to control dental plaque formation. More recently, the addition of nanoparticulate metals such as TiO2, SiO2, ZnO, Ag, CuO to dental materials to impart an antimicrobial effect, has been investigated in many studies. Among these metals, titanium dioxide nanoparticles have received the most attention due to its white color, low toxicity at concentrations usually used, high stability, availability, and its high photocatalytic activity.

Many studies suggested that incorporating titanium dioxide nanoparticles to PMMA, significantly decreases porosities in the denture resin, rendering titanium dioxide nanoparticles a suitable additive to denture base materials.

Titanium Dioxide as a Photocatalyst In 1977 Frank and Bard were the first to study the possibilities of using TiO2 to degrade cyanide in water, since then, there has been growing interest in its various applications.

Titanium dioxide is a light-sensitive semiconductor, that absorbs electromagnetic radiation in the near UV region. Absorbing light energy causes an electron to be promoted from the valence band to the conduction band.

Water molecules which are commonly adsorbed onto the titanium dioxide surface, are oxidized in the process, generating OH• radicals. These free radicals are characterized by a high level of energy enabling them to react with different organic compounds such as the polyunsaturated phospholipid component of the microbial lipid membrane that eventually leads to their complete oxidation to carbon dioxide and water, inhibiting the microorganisms' respiratory activity, and eliciting cell death.

Recent studies have proved the antimicrobial effects of titanium dioxide against Candida albicans, Staphylococcus aureus, Pseudomonas aeruginosa, Escherichia coli, Lactobacillus acidophilus, and MRSA.

However, there are recent concerns titanium dioxide could be cited as a health hazard, as it could produce tissue inflammation as generated by cytokine release. Moreover, adding TiO2 nanoparticles can alter the physical properties of the substrate. It has been found that adding as much as 5%wt of TiO2 nanoparticles to PMMA does not produce deleterious effects on the mechanical properties of the material, while concentrations required to produce an inhibitory or a killing effect on microorganisms has been found to be 0.25-2.5 mg/mL

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 40-70 years.
2. Completely edentulous participants.
3. Participants with well-developed ridges.
4. Compliant participants
5. Cooperative participants
6. Male or female participants

Exclusion Criteria:

1. Pathological changes of residual ridges.
2. Participants with any debilitating disease.
3. Participants with uncontrolled diabetes.
4. Participants with allergy to resins.
5. Participants with allergy to titanium dioxide nanoparticles.
6. Participants with severe undercuts, or irregular bony exostosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Bacterial Growth | 1 month
  Bacterial colony forming units